CLINICAL TRIAL: NCT01246843
Title: Evaluation of Cognitive Function of Patients Treated With Sunitinib or Sorafenib
Brief Title: Evaluation of Cognitive Function of Patients With Sunitinib or Sorafenib
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCNONCO200904
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Metastatic Renal Cell Cancer; GIST
Keywords: sunitinib; sorafenib; cognitive functioning
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- metastatic Renal Cell Carcinoma without treatment: patients with metastasized RCC who did not receive treatment
- mRCC with treatment: patients with metastastic renal cell cancer or GIST who are on treatment with Sunitinib or Sorafenib for
  ≥ 8 weeks

SUMMARY:
Patients with advanced kidney cancer or GIST (Gastro Intestinal Stromal Tumor: this is a tumor of the intestines) may be eligible for treatment with one of the following drugs: sunitinib (Sutent ®) or sorafenib (Nexavar ®). These drugs inhibit blood vessel formation in cancer cells. These cancer cells are hampered in their growth. To enlarge the investigators knowledge on the effects and side effects of these two medicines, in the University Medical Center St. Radboud lot of research is done. This study is a part of that.

Patients receiving sunitinib or sorafenib tell sometimes that they feel that they are less able to concentrate, that their memory is not working properly or that they are less able to imagine a solution to a complex problem . Perhaps you recognize these symptoms as well. In how many of the patients this occurs, how severe the symptoms are and how it is caused, is still unknown.

The goal of this research is to examine how memory, concentration and knowledge processing works in patients using sorafenib or sunitinib. With the research the investigators hope to get answers to the following questions:

1. How common are problems with memory, concentration and processing of knowledge in patients receiving the drug sunitinib or sorafenib?
2. What are the problems of memory, concentration and processing of knowledge in the use of sunitinib or sorafenib?
3. What could be the cause of the problems that patients experience from memory, concentration and processing of knowledge in the use of sunitinib or sorafenib?
4. Is there a link between problems with memory, concentration and processing of knowledge and also experiences of fatigue or mood of a patient?

DETAILED DESCRIPTION:
In this study we will focus on subjective and objective cognitive dysfunctioning in patients with metastatic cancer, treated with sunitinib or sorafenib. In our own clinical practice a substantial part of our patients that are treated with targeted therapies directed against VEGF, mention that they have problems with concentrating and that their memory function is decreased. Relatives sometimes point out that the behaviour of the patient is slightly different than before starting the VEGF (Vascular Endothelial Growth Factor) inhibition. Pre-clinical studies show that VEGF influences growth and recovery of neurons.

ELIGIBILITY:
Inclusion Criteria:

* Patients:
* patients with metastatic renal cell cancer or GIST who are on treatment with Sunitinib or Sorafenib for ≥ 8 weeks
* Karnofsky score > 70%
* age > 18 year.
* written informed consent for study

Patient controls selection

* patients with metastatic renal cell cancer or GIST who aren't treated yet (only interferon alfa or interleukine 2 treatment is allowed when > 12 months ago.
* Karnofsky score > 70%
* age > 18 year.
* written informed consent for study

Exclusion Criteria:

* Patients:
* contra-indications for treatment with Sunitinib or Sorafenib
* patients who do not speak or write the Dutch language adequately
* known brain metastasis
* use of psychiatric or anti-epileptic medication
* known cognitive disorders unrelated to diagnosis or medication use
* radiotherapy on the brain at any time in the past
* systemic chemotherapy
* in the last 12 months interferon alfa or interleukin-2 treatment
* operation in the last 3 months
* Stroke/TIA (transient ischaemic attack)

Patient controls section:

* patients who do not speak or write the Dutch language adequately
* known brain metastasis
* use of psychiatric or anti-epileptic medication
* known cognitive disorders unrelated to diagnosis or medication use
* radiotherapy on the brain at any time in the past
* systemic chemotherapy
* in the last 12 months interferon alfa or interleukin-2 treatment
* operation in the last 3 months
* stroke/TIA (transient ischaemic attack)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mRCC are asked by their own physician.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, Md PhD, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Mulder SF, Bertens D, Desar IM, Vissers KC, Mulders PF, Punt CJ, van Spronsen DJ, Langenhuijsen JF, Kessels RP, van Herpen CM. Impairment of cognitive functioning during Sunitinib or Sorafenib treatment in cancer patients: a cross sectional study. BMC Cancer. 2014 Mar 24;14:219. doi: 10.1186/1471-2407-14-219. PMID 24661373